CLINICAL TRIAL: NCT01277302
Title: A Multicenter Randomized Study Evaluating Dosing Regimens for Treatment With Intravitreal Ranibizumab Injections in Subjects With Macular Edema Following Retinal Vein Occlusion
Brief Title: A Study Evaluating Dosing Regimens for Treatment With Intravitreal Ranibizumab Injections in Subjects With Macular Edema Following Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4967g; ML01296 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

ARMS (3):
- Ranibizumab 0.5 mg monthly - randomized subjects (Experimental): Subjects received at least 7 monthly intravitreal ranibizumab 0.5 mg injections until the first month where the study-specific visual acuity and spectral-domain optical coherence tomography (VA-OCT) stability criteria were met and randomization occurred to the monthly arm. At subsequent monthly visits after randomization, injections were given whether the VA-OCT stability criteria were met or not met. Subjects were to receive 15 ranibizumab 0.5 mg injections.
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.5 mg PRN - randomized subjects (Experimental): Subjects received at least 7 monthly intravitreal ranibizumab 0.5 mg injections until the first month where the study-specific VA-OCT stability criteria were met and randomization occurred to the PRN arm. No injection was given at the randomization visit. At subsequent monthly visits after randomization, injections were given if the VA-OCT stability criteria were not met and no injections were given if the VA-OCT stability criteria were met. Subjects could receive between 7 and a maximum of 14 ranibizumab 0.5 mg injections.
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.5 mg monthly - non-randomized subjects (Experimental): Subjects received at least 7 monthly intravitreal ranibizumab 0.5 mg injections and then never met the study-specific VA-OCT stability criteria from month 7 to month 14. Subjects were to receive 15 ranibizumab 0.5 mg injections.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Liquid ranibizumab (10 mg/ml) was supplied in a sterile solution in single-use vials.
  Other Names: Lucentis

SUMMARY:
This was a Phase IV multicenter, randomized, open-label study, with masking of the vision examiner, of the efficacy and safety of intravitreal ranibizumab 0.5 mg in subjects with macular edema following Branch Retinal Vein Occlusion (BRVO) or Central Retinal Vein Occlusion (CRVO).

DETAILED DESCRIPTION:
This study consisted of 2 study periods, a 7-month fixed treatment period, followed by an 8-month alternate dose regimen period. Subjects could receive up to a maximum of 15 monthly injections of ranibizumab 0.5 mg during the study, 7 injections (Day 0 and at 6 monthly visits) in the fixed treatment period and a maximum of 8 injections in the alternate dose regimen period. During the fixed treatment period, subjects received 7 monthly intravitreal ranibizumab 0.5 mg injections. During the alternate dose regimen period, from Month 7 through Month 14, subjects were evaluated monthly to determine whether they achieved the study-specific visual acuity and spectral-domain optical coherence tomography (VA-OCT) stability criteria. Subjects continued to receive monthly ranibizumab 0.5 mg monthly injections until the VA-OCT stability criteria were first met. Upon meeting the VA-OCT stability criteria for the first time during the alternate dose regimen period, subjects were randomly assigned in a 1:1 ratio to one of 2 dose regimens, the PRN (pro re nata, "as-needed") or the Monthly regimen.

PRN randomized subjects: Subjects received no injection at the randomization visit and at future monthly visits where the VA-OCT stability criteria were met and received a ranibizumab 0.5 mg injection at future monthly visits if the VA-OCT stability criteria were not met.

Monthly randomized subjects: Subjects continued to receive ranibizumab 0.5 mg injections at each monthly visit.

Monthly non-randomized subjects: Subjects who did not meet the VA-OCT stability criteria at any month from Month 7 through Month 14 were not randomized and received 8 monthly intravitreal ranibizumab 0.5 mg injections.

ELIGIBILITY:
Inclusion Criteria:

* For sexually active women of childbearing potential, use of an appropriate form of contraception (or abstinence) for the duration of the study.

Ocular Inclusion Criteria (Study Eye)

* Foveal center-involved macular edema secondary to branch retinal vein occlusion (BRVO) (including hemi-retinal retinal vein occlusion [HRVO]) or central retinal vein occlusion (CRVO).
* Best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) charts of 20/40 to 20/320 (Snellen equivalent) in the study eye.
* Mean central subfield thickness > 300 µm on 2 spectral-domain optical coherence tomography measurements (screening and Day 0 [first day of treatment]).

Exclusion Criteria:

* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.
* History of any systemic anti-vascular endothelial growth factor (VEGF) or pro-VEGF treatment within 6 months prior to Day 0.
* History of allergy to fluorescein.
* History of allergy to ranibizumab injection or related molecule.
* Relevant systemic disease that may be associated with increased systemic VEGF levels. History of successfully treated malignancies is not an exclusion criterion.
* Uncontrolled blood pressure.
* Pregnancy or lactation.
* Daily use of oral corticosteroids to treat a chronic condition.
* Required treatment with injectable corticosteroids to treat a musculoskeletal condition.
* Participation in an investigational trial within 30 days prior to Day 0 that involved treatment with any drug or device that has not received regulatory approval at the time of study entry.

Ocular Exclusion Criteria (Study Eye)

* Prior episode of retinal vein occlusion (RVO).
* Brisk afferent pupillary defect.
* History of any previous intravitreal anti-VEGF therapy for RVO in the study eye.
* History of previous therapeutic treatment for RVO, other than anti-VEGF therapy, within 4 months prior to the screening visit, including any intraocular corticosteroids.
* History of previous surgical treatment for RVO, including radial optic neurotomy or sheathotomy.
* History or presence of age-related macular degeneration (AMD) (dry form graded as Age-Related Eye Disease Study [AREDS] Stage 2 or higher or wet form).
* History of laser photocoagulation for macular edema within 4 months prior to Day 0.
* History of panretinal scatter photocoagulation or sector laser photocoagulation within 4 months prior to Day 0 or anticipated within the next 4 months following Day 0.
* History of pars plana vitrectomy.
* History of intraocular surgery within 2 months prior to Day 0 or anticipated within the next 7 months following Day 0.
* History of yttrium-aluminum-garnet (YAG) capsulotomy performed within 2 months prior to Day 0.
* Previous filtration surgery in the study eye.
* History of herpetic ocular infection.
* History of ocular toxoplasmosis.
* History of rhegmatogenous retinal detachment.
* History of idiopathic central serous chorioretinopathy.
* Evidence upon examination of vitreoretinal interface disease either on clinical examination or spectral-domain optical coherence tomography (SD-OCT), thought to be contributing to macular edema.
* Presence of an ocular condition that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the study.
* Visually significant hemorrhage obscuring the fovea and felt to be a major contributor to reduced visual acuity. The subject should be followed and when the hemorrhage in the fovea clears to the point that it is no longer a major contributor to reduced visual acuity, the subject may be screened for the study.
* Presence of a substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more.
* Intra-ocular pressure (IOP) ≥ 30 mmHg. If a subject's IOP is ≥ 30 mmHg, that subject will be referred for glaucoma treatment and may be re-screened after 1 month.
* Evidence upon examination of pseudoexfoliation.
* Aphakia.
* Evidence upon examination of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.
* Evidence upon examination of any diabetic retinopathy, defined as eyes of diabetic patients with more than one microaneurysm outside the area of the vein occlusion (inclusive of both eyes).
* Other relevant ocular disease that may be associated with increased intraocular VEGF levels.
* Improvement of ≥ 10 letters on best-corrected visual acuity ETDRS score between screening and Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Sternberg, M.D., Study Director — Genentech, Inc.
Locations (41):
- United States (41):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Chico, California
  - Mountain View, California
  - Oakland, California
  - San Francisco, California
  - Santa Ana, California
  - Santa Barbara, California
  - Torrance, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Lakeland, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Jackson, Michigan
  - Edina, Minnesota
  - Las Vegas, Nevada
  - Northfield, New Jersey
  - Teaneck, New Jersey
  - Rochester, New York
  - Charlotte, North Carolina
  - Camp Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas

REFERENCES:
- [Derived] Yiu G, Huang D, Wang Y, Wang Z, Yang M, Haskova Z. Predictors of As-Needed Ranibizumab Injection Frequency in Patients With Macular Edema Following Retinal Vein Occlusion. Am J Ophthalmol. 2023 May;249:74-81. doi: 10.1016/j.ajo.2023.01.004. Epub 2023 Jan 14. PMID 36646240
- [Derived] Lloyd Clark W, Liu M, Kitchens J, Wang PW, Haskova Z. Baseline characteristics associated with early visual acuity gains after ranibizumab treatment for retinal vein occlusion. BMC Ophthalmol. 2019 Jan 8;19(1):11. doi: 10.1186/s12886-018-1012-y. PMID 30621653

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab 0.5 mg PRN - Randomized Subjects: Subjects received at least 7 monthly intravitreal ranibizumab 0.5 mg injections until the first month where the study-specific VA-OCT stability criteria were met and randomization occurred to the PRN arm and no injection was given. At subsequent monthly visits after randomization, injections were given if the VA-OCT stability criteria were not met and no injections were given if the VA-OCT stability criteria were met. Subjects could receive between 7 and a maximum of 14 ranibizumab 0.5 mg injections.
Period: 7-Month Fixed Treatment Period
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Started | 85 | 86 | 31
Completed | 85 | 86 | 19
Not Completed | 0 | 0 | 12
Not completed — Subject Decision to Withdraw | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Subject Required Other Drug Therapy | 0 | 0 | 1
Not completed — Subject Non-compliance | 0 | 0 | 1
Period: 8-Month Alternate Dose Regimen Period
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Started | 85 | 86 | 19
Completed | 80 | 82 | 13
Not Completed | 5 | 4 | 6
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Subject Decision to Withdraw | 3 | 0 | 1
Not completed — Subject Non-compliance | 0 | 2 | 1
Not completed — Relocation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All enrolled participants who received at least 1 ranibizumab injection in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects | Total
Number analyzed (Participants) | 85 | 86 | 31 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (12.1) | 65.2 (12.8) | 66.3 (12.3) | 66.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 9 | 84
  Male | 47 | 49 | 22 | 118

OUTCOME MEASURES:

1. Primary Outcome: Trend of Change From Baseline in the Best Corrected Visual Acuity (BCVA) Scores From Month 7 to Month 15
Description: BCVA was measured in the study eye using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision. A positive change score indicates improvement. The reported data are the observed changes from Baseline in BCVA at Months 7 and 15. For the statistical analysis, the interaction term of treatment by time in a longitudinal model was used to assess whether there was a difference in the trend of change from Baseline in the visual acuity scores from Month 7 to Month 15 between the 2 randomized treatment groups, Monthly and PRN.
Time Frame: Baseline to Month 15
Population: Intent-to-treat population, randomized: All enrolled participants who received at least 1 ranibizumab injection in the study and were randomized into the Monthly or PRN treatment groups. The analysis was based on observed data without imputation for missing values.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects
Number analyzed (Participants) | 85 | 86
Letters
  Month 7 (n=85, 86) | 17.5 (12.6) | 19.7 (12.6)
  Month 15 (n=80, 82) | 18.7 (14.1) | 21.0 (14.1)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg Monthly - Randomized Subjects vs Ranibizumab 0.5 mg PRN - Randomized Subjects; The null hypothesis was that there was no difference in the trend of change from Baseline in the visual acuity scores from Month 7 to Month 15 between the 2 treatment groups as assessed by the interaction term of treatment by time in a longitudinal model; Test type: Superiority or Other; p = 0.5091, Longitudinal mixed model — This is the p-value of the treatment by time interaction in the longitudinal model. Analysis was not adjusted for multiple comparisons as there was only 1 comparison. p < 0.05 (2-sided) was required for significance; The analysis was stratified by disease (BRVO or CRVO), randomization month, and randomization BCVA score category (≤35, >35 to ≤50, or >50 letters); Estimated interaction effect = 0.071, Standard Error of Mean 0.107

2. Secondary Outcome: Visual Acuity Change From Previous Month During the Alternate Dose Regimen Period in Subjects Who Met the VA-OCT Stability Criteria at the Previous Month
Description: BCVA was measured in the study eye using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision. A positive change score indicates improvement. This outcome measure is not relevant for subjects in the non-randomized group because they never met the VA-OCT stability criteria.
Time Frame: Month 7 through Month 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects
Number analyzed (Participants) | 85 | 86
Letters
  Month 8 (n=53, 53) | 0.4 (3.2) | -3.3 (11.3)
  Month 9 (n=49, 40) | 0.5 (4.0) | -2.9 (8.6)
  Month 10 (n=52, 31) | 0.2 (3.4) | -0.5 (4.2)
  Month 11 (n=54, 40) | -0.6 (3.7) | 0.4 (4.4)
  Month 12 (n=46, 44) | -0.2 (3.2) | -1.6 (4.4)
  Month 13 (n=50, 41) | 0.0 (3.5) | -0.5 (5.2)
  Month 14 (n=58, 48) | -0.1 (3.6) | -2.2 (6.1)
  Month 15 (n=56, 42) | 0.0 (4.4) | -0.4 (4.0)

3. Secondary Outcome: Percentage of Participants Who Gained ≥ 15 Letters in Their Best Corrected Visual Acuity (BCVA) Score From Baseline
Description: BCVA was measured in the study eye using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision.
Time Frame: Month 7 to Month 15
Population: Intent-to-treat population: All enrolled participants who received at least 1 ranibizumab injection in the study. The analysis was based on observed data without imputation for missing values.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
Percentage of participants
  Month 7 (n=85, 86, 17) | 62.4 [52.1 to 72.7] | 67.4 [57.5 to 77.3] | 41.2 [17.8 to 64.6]
  Month 15 (n=80, 82, 13) | 66.3 [55.9 to 76.6] | 70.7 [60.9 to 80.6] | 46.2 [19.1 to 73.3]

4. Secondary Outcome: Percentage of Participants With a Visual Acuity (VA) Snellen Equivalent of 20/40 or Better
Description: VA was measured in the study eye using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart starting at a test distance of 4 meters. An increase in the number of lines read correctly by the patient in the ETDRS chart indicates an improvement of vision. The Snellen equivalent of 20/40 or better is 69 or more letters correctly read in the EDTRS chart.
Time Frame: Month 7 to Month 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
Percentage of participants
  Month 7 (n=85, 86, 17) | 72.9 [63.5 to 82.4] | 76.7 [67.8 to 85.7] | 47.1 [23.3 to 70.8]
  Month 15 (n=80, 82, 13) | 71.3 [61.3 to 81.2] | 76.8 [67.7 to 86.0] | 46.2 [19.1 to 73.3]

5. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Score
Description: BCVA was measured in the study eye using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient. An increase in the BCVA score indicates an improvement of vision. A positive change score indicates improvement.
Time Frame: Month 1 to Month 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
Letters
  Month 1 (n=85, 86, 29) | 12.2 (10.3) | 11.2 (10.4) | 10.7 (14.0)
  Month 7 (n=85, 86, 17) | 17.5 (12.6) | 19.7 (12.6) | 14.7 (12.0)
  Month 15 (n=80, 82, 13) | 18.7 (14.1) | 21.0 (14.1) | 14.5 (14.7)

6. Secondary Outcome: Percentage of Participants Who Lost < 15 Letters in Their Best Corrected Visual Acuity (BCVA) Score From Baseline
Description: as for outcome 3
Time Frame: Month 7 to Month 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
Percentage of participants
  Month 7 (n=85, 86, 17) | 98.8 [96.5 to 100.0] | 98.8 [96.6 to 100.0] | 100.0 [NA to NA] — A 95% confidence interval cannot be calculated for the observed percentage of 100%.
  Month 15 (n=80, 82, 13) | 98.8 [96.3 to 100.0] | 98.8 [96.4 to 100.0] | 100.0 [NA to NA] — A 95% confidence interval cannot be calculated for the observed percentage of 100%.

7. Secondary Outcome: Percentage of Participants With a Central Foveal Thickness of ≤ 300 µm
Description: Central foveal thickness was assessed monthly in the study eye using spectral-domain optical coherence tomography. Central foveal thickness was computed using the automated Cirrus Review software (DOCTR CZM Cirrus OCT Grader Reading Manual, Version 1.02). All participants in the Monthly and PRN groups had a baseline central foveal thickness > 300 µm at baseline.
Time Frame: Month 7 to Month 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
Percentage of participants
  Month 7 (n=85, 86, 17) | 88.2 [81.4 to 95.1] | 94.2 [89.2 to 99.1] | 52.9 [29.2 to 76.7]
  Month 15 (n=80, 82, 13) | 92.5 [86.7 to 98.3] | 85.4 [77.7 to 93.0] | 38.5 [12.0 to 64.9]

8. Secondary Outcome: Mean Change From Baseline in Central Foveal Thickness
Description: Central foveal thickness was assessed monthly in the study eye using spectral-domain optical coherence tomography. Central foveal thickness was computed using the automated Cirrus Review software (DOCTR CZM Cirrus OCT Grader Reading Manual, Version 1.02). All participants in the Monthly and PRN groups had a baseline central foveal thickness > 300 µm at baseline. A decrease in foveal thickness suggests a reduction in macular edema. A negative change score indicates improvement.
Time Frame: Month 1 to Month 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
µm
  Month 1 (n=85, 86, 29) | -243.0 (172.5) | -214.9 (166.7) | -157.9 (181.8)
  Month 7 (n=85, 86, 17) | -279.7 (167.4) | -265.2 (185.9) | -113.9 (184.9)
  Month 15 (n=80, 82, 13) | -289.9 (177.2) | -247.8 (207.5) | -93.2 (225.2)

9. Secondary Outcome: Percentage of Participants With Intraretinal Edema
Description: The presence of intraretinal edema was defined as the presence of subretinal fluid, cystoid spaces, or central retinal thickness ≥ 300 µm as evaluated in spectral-domain optical coherence tomography images by the Digital Angiography Reading Center, the central reading center. At baseline, all participants in the Monthly and PRN groups had presence of edema.
Time Frame: Month 7 to Month 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Number analyzed (Participants) | 85 | 86 | 31
Percentage of participants
  Month 7 (n=85, 86, 17) | 31.8 [21.9 to 41.7] | 30.2 [20.5 to 39.9] | 100.0 [NA to NA] — A 95% confidence interval cannot be calculated for the observed percentage of 100%.
  Month 15 (n=80, 82, 13) | 25.0 [15.5 to 34.5] | 32.9 [22.8 to 43.1] | 84.6 [65.0 to 100.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were reported beginning at initiation of study treatment up to 30 days following the last administration of study treatment, study discontinuation, or termination, whichever was earlier.
Description: After this period, only SAEs attributed to prior study treatment were reported. Safety population: All enrolled participants who received at least 1 ranibizumab injection in the study.
Arm/Group | Ranibizumab 0.5 mg Monthly - Randomized Subjects | Ranibizumab 0.5 mg PRN - Randomized Subjects | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects
Serious Adverse Events (participants affected / at risk) | 12/85 | 14/86 | 11/31
Other Adverse Events (participants affected / at risk) | 70/85 | 61/86 | 18/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg Monthly - Randomized Subjects (N=85) | Ranibizumab 0.5 mg PRN - Randomized Subjects (N=86) | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Non-cardia chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 0 | 1 — Study eye
Macular oedema (Eye disorders) | 0 | 0 | 1 — Study eye
Visual acuity reduced (Eye disorders) | 1 | 3 | 0 — Study eye
Iridocyclitis (Eye disorders) | 0 | 0 | 1 — Fellow eye
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 — Fellow eye
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg Monthly - Randomized Subjects (N=85) | Ranibizumab 0.5 mg PRN - Randomized Subjects (N=86) | Ranibizumab 0.5 mg Monthly - Non-randomized Subjects (N=31)
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Bronchitis (Infections and infestations) | 4 | 3 | 2
Nasopharyngitis (Infections and infestations) | 10 | 7 | 1
Sinusitis (Infections and infestations) | 3 | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 6 | 0
Blood pressure increased (Investigations) | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 13 | 8 | 2
Cataract (Eye disorders) | 9 | 6 | 0 — Study eye
Cataract cortical (Eye disorders) | 4 | 5 | 1 — Study eye
Conjunctival haemorrhage (Eye disorders) | 28 | 23 | 9 — Study eye
Dry eye (Eye disorders) | 4 | 3 | 2 — Study eye
Eye irritation (Eye disorders) | 6 | 5 | 1 — Study eye
Eye pain (Eye disorders) | 8 | 14 | 4 — Study eye
Eye pruritus (Eye disorders) | 1 | 4 | 2 — Study eye
Macular fibrosis (Eye disorders) | 9 | 5 | 2 — Study eye
Macular hole (Eye disorders) | 1 | 0 | 2 — Study eye
Macular oedema (Eye disorders) | 2 | 6 | 1 — Study eye
Retinal aneurysm (Eye disorders) | 1 | 5 | 0 — Study eye
Retinal depigmentation (Eye disorders) | 2 | 0 | 2 — Study eye
Retinal disorder (Eye disorders) | 7 | 1 | 1 — Study eye
Retinal exudates (Eye disorders) | 13 | 12 | 3 — Study eye
Retinal haemorrhage (Eye disorders) | 8 | 8 | 0 — Study eye
Retinal vascular disorder (Eye disorders) | 3 | 5 | 0 — Study eye
Vitreous adhesions (Eye disorders) | 0 | 0 | 3 — Study eye
Vitreous detachment (Eye disorders) | 11 | 6 | 3 — Study eye
Vitreous floaters (Eye disorders) | 4 | 6 | 1 — Study eye
Intraocular pressure increased (Investigations) | 3 | 8 | 1 — Study eye
Cataract (Eye disorders) | 8 | 5 | 0 — Fellow eye
Dry eye (Eye disorders) | 3 | 2 | 2 — Fellow eye
Retinal haemorrhage (Eye disorders) | 4 | 6 | 0 — Fellow eye
Vitreous detachment (Eye disorders) | 7 | 2 | 1 — Fellow eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.